CLINICAL TRIAL: NCT02821676
Title: A Randomized Controlled Comparison of PECI/SPB Versus Intercostal Nerve Block for the Management of Postoperative Pain in Latissimus Dorsi Flap Reconstruction
Brief Title: PECI/SPB vs Intercostal Nerve Block for the Management of Postoperative Pain in Latissimus Dorsi Flap Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Jing Zhang, Staff Plastic Surgeon, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20160235-01H
Record Dates: First submitted 2016-05-31; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEC1/SPB Block (Experimental)
  Interventions: Procedure: PECI/SPB Block with Active Anesthetic + Placebo Multilevel Intercostal Nerve Block followed by Latissimus Dorsi Flap Breast Reconstruction
- Intercostal Block (Active Comparator)
  Interventions: Procedure: Placebo PEC/SPB Block + Multilevel Intercostal Nerve Block with Active Anesthetic followed by Latissimus Dorsi Flap Breast Reconstruction

INTERVENTIONS:
Procedure: PECI/SPB Block with Active Anesthetic + Placebo Multilevel Intercostal Nerve Block followed by Latissimus Dorsi Flap Breast Reconstruction — 30mL of 0.5% Ropivacaine with 1:200,000 epinephrine preoperatively via an ultrasound guided PECI/SPB regional block and 5mL of Normal Saline intraoperatively as an intercostal nerve block to each of the T2-T7 nerve segments
  Arms: PEC1/SPB Block
Procedure: Placebo PEC/SPB Block + Multilevel Intercostal Nerve Block with Active Anesthetic followed by Latissimus Dorsi Flap Breast Reconstruction — 30mL of Normal Saline via an ultrasound guided PECI/SPB block and 5mL of 0.5% Ropivacaine with 1:200,000 epinephrine as an Intercostal nerve block to each of the T2-T7 nerve segments
  Arms: Intercostal Block

SUMMARY:
Regional Anesthesia is a procedure in which numbing medication is injected around nerves that transmit pain from areas involved in a surgery. The objective is to block the nerves so a patient does not feel pain after surgery. Regional nerve blocks offer many advantages over traditional anesthetic techniques, including faster recovery time, fewer side effects and a dramatic reduction in post-surgical pain.

The use of regional anesthesia in breast reconstructive surgery, such as the latissimus dorsi flap, has led to major improvements in patient care. Today, the most common regional anesthetic used in latissimus dorsi flap reconstruction is the intercostal nerve block, where numbing medication is injected around the nerves supplying the chest wall.

While intercostal nerve blocks have been used successfully in breast surgery, they do not provide a complete nerve block to the chest wall, as there are some nerves that are unaccounted for in the block which can contribute to a patients pain after surgery.

The mixed pectoral one / serratus plane block (PECI/SPB) block is another regional nerve block that has been successfully used by anesthesiologists at The Ottawa Hospital and offers a more complete pain blockade than the intercostal nerve block, as it includes more nerves that supply the breast. In addition to this, the intercostal nerve block is a so-called "blind-technique" compared to the PECI/SPB block, which is more accurately guided by ultrasound. Blind techniques are associated with higher failure rates.

Both the intercostal nerve block and the PECI/SPB nerve block have been used successfully at the Ottawa Hospital. In this study, the investigators propose a prospective, double blinded, randomized controlled, head to head comparison of the PECI/SPB and intercostal nerve block to determine which block is associated with the best pain blockade and patient satisfaction in lattissimus dorsi flap surgery.

DETAILED DESCRIPTION:
Recent literature has unequivocally demonstrated that postoperative pain remains under-treated in hospitals. While breast surgery remains one of the most common surgeries performed in hospitals today, it has been shown that 40% of women still experience meaningful pain postoperatively. It is well known that poor pain control is not only associated with slower recovery, longer admission in hospital and poor patient satisfaction but it also can lead to the development of chronic post surgical pain.

In recent years, regional nerve blocks have emerged as a promising adjunct to standard postoperative analgesic ladder protocols. The main advantage of regional anesthesia is the reduction of postoperative pain while limiting the amount of oral and intravenous narcotic use. The reduction of postoperative narcotic use is advantageous for the patient and caregiver alike as it reduces common side effects associated with such medications, such as drowsiness, nausea, vomiting, upset stomach and dizziness.

Regional anesthesia in breast reconstruction surgery commonly include thoracic epidurals, intercostal nerve blocks and paravertebal nerve blocks. To date, there remains no standard of care for perioperative pain management and it is usually left to the discretion of the surgeon and anesthesiologist involved to decide which pain blockade is preferable on a case by case basis. While paravertebral and intercostal nerve blocks have shown promising results, they do not provide a complete sensory block to the anterior chest wall, as innervation is supplied not only from the thoracic spinal nerves but also via medial and lateral pectoral nerves off the brachial plexus.

The pectoral nerve block is a novel interfascial block placed into the plane between pectoralis major and minor muscles and is particularly useful in reconstructive breast surgery involving subpectoral prosthesis. It has been associated with minimal analgesia postoperatively and is thought to be particularly useful in the daycare setting.

To the best of the knowledge of the investigators, the utility of the pectoral nerve block in pedicled Latissimus Dorsi breast reconstruction has not been investigated. A mixed PEC I/ Serratus Plane Block provides analgesia to the lateral and medial pectoral nerves, lateral and anterior branches of the T2-T4 spinal nerves, long thoracic nerve and thoracodorsal nerve, theoretically offering a more comprehensive block than the midaxillary intercostal block and with no additional morbidity to the patient. Furthermore, the intercostal nerve block is a blind technique that may be associated with higher failure rates compared to the more precise, ultrasound guided, PECI/SPB block.

In this study, the investigators plan to systematically investigate these two blocks in latissimus dorsi flap reconstruction in order to document optimal postoperative pain management.

ELIGIBILITY:
Inclusion Criteria:

* Breast Reconstruction using the Latissimus Dorsi Flap

Exclusion Criteria:

* All patients undergoing breast reconstruction using techniques other than the pedicled latissimus dorsi myocutaneous flap
* Preexisting diagnosis of a chronic pain disorder
* BMI > or = to 35/kg/m2
* History of allergy or sensitivity to local anesthetic
* History of coagulopathy or bleeding disorder
* Weight <50Kg
* Allergies to local anesthetic, celecoxib, acetaminophen, hydromorphone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Total 24 Hour Narcotic Usage | 24 hours
  This is the most common primary outcome used in the regional anesthesia literature when comparing nerve blocks.

SECONDARY OUTCOMES:
Time to first analgesic request (TFA) | 24 hours
Postoperative Pain score at 0h, 1h, 3h, 5h, 24 hours | 24 hours
Patient self reported pain score at 24 hours post-surgery | 24 hours
Peak expiratory flow rate | 24 hours
Breast Q Questionnaire | 24 hours
  Physical and Psychological well-being questionnaire after breast reconstruction
QoR-40 Patient Satisfaction Questionnaire | 24 hours
  Perioperative Care Satisfaction Questionnaire

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will not be made available. Anonymity will be maintained throughout the study.